CLINICAL TRIAL: NCT03114150
Title: Exercise to Improve Hippocampal Connectivity and Learning in Older Adults
Brief Title: Exercise Effects on Brain Health and Learning From Minutes to Months
Acronym: EXTEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle W. Voss (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Michelle W. Voss, Associate Professor of Psychological and Brain Sciences, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 201705800; 1R01AG055500-01 (NIH)
Record Dates: First submitted 2017-03-30; First posted 2017-04-14 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Sedentary Lifestyle
Keywords: physical activity; aging; learning and memory; exercise; brain
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiorespiratory fitness training (Experimental): Cardiorespiratory fitness training will be a 24-week supervised cycling program designed to improve cardiorespiratory fitness, with supervision directly from the research team. All participants will first receive a one-on-one orientation with an exercise training specialist that has been trained by Dr. Gary Pierce in monitoring an exercise program for healthy older adults. Training will start with a 5 minute-warm-up, 20 minutes moderate intensity cycling and 30 minutes light intensity cycling, and 5 minute cool-down per session, for 3 sessions/week. In each additional week, 6 minutes of moderate intensity cycling per session will be added, until the total time for moderate intensity is 50 minutes per session by the start of week 5 (with additional 5 minute warm-up and 5 minute cool-down).
  Interventions: Behavioral: Cardiorespiratory fitness training
- Functional fitness training (Active Comparator): Functional fitness training will be a 24-week supervised exercise program designed to focus on functional flexibility and mobility, with supervision directly from our research team. All participants will first receive a one-on-one orientation with an exercise training specialist that has been trained by Dr. Gary Pierce in monitoring an exercise program for healthy older adults. Training will start with a 5 minute-warm-up, 20 minutes of light intensity cycling and 20 minutes of dynamic stretching to increase range of motion and functional fitness, for 3 sessions/week. In each additional week, additional stretches will be added to maintain variety and improve flexibility of all major muscle groups.
  Interventions: Behavioral: Functional fitness training

INTERVENTIONS:
Behavioral: Cardiorespiratory fitness training — Physical exercise of moderate intensity designed to improve cardiorespiratory fitness
  Arms: Cardiorespiratory fitness training
Behavioral: Functional fitness training — Physical exercise of light intensity designed to improve functional fitness
  Arms: Functional fitness training

SUMMARY:
Given the accelerating growth of older adults worldwide and the decline in cognitive function with aging, therapeutics that remediate age-related cognitive decline are needed more than ever. The proposed research seeks to better understand and enhance the detection of exercise effects on hippocampal network function and learning and memory, which decline with aging and Alzheimer's. Success would lead to new ways to detect benefits of exercise on cognitive aging and would lead to mechanistic insight on how such plasticity is possible while also informing prevention strategies.

DETAILED DESCRIPTION:
Animal models robustly support that exercise protects brain areas vulnerable to aging such as the hippocampus and that these benefits lead to better learning. In contrast, there are mixed findings from human studies on the cognitive benefits of exercise with healthy older adults. This contrast indicates there is still a lack of understanding for how exercise could change the course of cognitive decline in aging adults. However, no human studies have comprehensively tested exercise effects on cognition in older adults with learning tasks inspired from basic exercise neuroscience. The objective in the proposed research is to fill this translational gap by determining if different types of exercise improve the same kinds of learning in older adults that have been shown to improve in animal models by improving hippocampal function. This will bring the investigators closer to a long-term goal of determining how exercise protects the brain from adverse effects of aging in order to develop interventions that minimize age-related cognitive decline. The overall hypothesis is that exercise improves learning when it increases functional hippocampal-cortical communication that otherwise declines with aging. The investigators will test this in a sample of healthy older adults by determining if increases in functional hippocampal-cortical connectivity from exercise training improve learning on an array of tasks that require the hippocampus for acquisition of new relational memories compared to conditions of the same tasks that should not require the hippocampus for learning and memory.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to participate in an aerobic exercise intervention based on the Physical Activity Readiness Questionnaire, and corrected vision of 20/40.
* Approval from a physician that monitored electrocardiography (ECG) response during a maximal aerobic fitness test that is part of the second study visit described below.
* Exercising less than 60 minutes a week for the past calendar year

Exclusion Criteria:

* Not between the ages of 55 and 80 years old
* Not fluent in English
* Score < 20 (out of 30) on the Montreal Cognitive Assessment (MoCA)
* Inability to comply with experimental instructions
* Qualify as "high risk" for acute cardiovascular event by the published standards of the American College of Sports Medicine
* Previous diagnosis of neurological, metabolic, or psychiatric condition, and no previous brain injury associated with loss of consciousness
* Inability to complete an MRI

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle W Voss, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
In accord with NIH regulations, the investigators will make the data and relevant documentation available to other investigators upon acceptance of the main findings from the study for publication. The investigators will share analysis tools as they are developed. Because the collected data are to remain anonymous, only a subject number will identify all data. To further protect the privacy and confidentiality of the data, data and documentation will be made available only under a data-sharing agreement that provides for restrictions for the transferring of data to others and a commitment that the data will be used for research purposes only and not for a profit-making enterprise.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We will share baseline neuroimaging data and phenotypic data upon completion of data collection. We will share the intervention outcome data after we have published our results from each primary aim.
Access Criteria: We will share on an open platform such as OpenNeuro (https://openneuro.org/).

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate Intensity Aerobic Exercise First, Then Light Intensity Aerobic Exercise: Crossover of Moderate Intensity Aerobic exercise condition followed by Light Intensity Aerobic Exercise for Acute exercise manipulation
- Light Intensity Aerobic Exercise First, Then Moderate Intensity Aerobic Exercise: Crossover of Light Intensity Aerobic exercise condition followed by Moderate Intensity Aerobic Exercise for Acute exercise manipulation
Period: Crossover: One Week
Arm/Group | Moderate Intensity Aerobic Exercise First, Then Light Intensity Aerobic Exercise | Light Intensity Aerobic Exercise First, Then Moderate Intensity Aerobic Exercise | Cardiorespiratory Fitness Training | Functional Fitness Training
Started | 58 | 64 | 0 | 0
Completed | 58 | 61 | 0 | 0
Not Completed | 0 | 3 | 0 | 0
Period: Randomized Trial: 24 Weeks
Arm/Group | Moderate Intensity Aerobic Exercise First, Then Light Intensity Aerobic Exercise | Light Intensity Aerobic Exercise First, Then Moderate Intensity Aerobic Exercise | Cardiorespiratory Fitness Training | Functional Fitness Training
Started | 0 | 0 | 60 | 56
Completed | 0 | 0 | 55 | 52
Not Completed | 0 | 0 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardiorespiratory Fitness Training | Functional Fitness Training | Total
Number analyzed (Participants) | 60 | 56 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (6) | 63.4 (5) | 63.3 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 35 | 76
  Male | 19 | 21 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 57 | 52 | 109
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 56 | 116
Cardiorespiratory fitness (VO2 max as ml/kg/min) [Mean (Standard Deviation); unit: VO2 max (ml/kg/min)] — Participants completed a symptom-limited maximal exercise test to exhaustion on an upright cycle ergometer with 12-lead electrocardiography (ECG) and cardiopulmonary gas analysis (True One, Parvomedics, Inc.) for determining VO2max supervised by a trained exercise specialist and licensed healthcare practitioner (cardiologist).
  VO2 max (ml/kg/min) | 20.1 (5.2) | 21.1 (5.8) | 20.6 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hippocampal-dependent Learning
Description: Learning rate on constructs that have been examined in animal models including context acquisition, episodic associations, and spatial navigation. The primary outcome is reported for the spatial navigation task that is associated with hippocampal structure and function, which is learning in the wayfinding condition. We report change in slope for wayfinding learning trials. The slope is computed based on the proportion of items correctly recalled on a map, over four learning trials. For each trial, proportion correct can range from 0 to 1, and a higher number represents faster learning, which is better.
Time Frame: Baseline, 24-weeks
Population: Participants with both pre- and post-intervention measurements.
Measure: Mean (Standard Deviation); unit: learning rate (proportion correct/trial)
Arm/Group | Cardiorespiratory Fitness Training | Functional Fitness Training
Number analyzed (Participants) | 48 | 45
learning rate (proportion correct/trial) | -.00369 (.03) | .00404 (.04)
Statistical Analysis 1: Comparison: Cardiorespiratory Fitness Training vs Functional Fitness Training; We tested the prediction that learning rate would increase more so for the moderate-to-vigorous training group compared to the light intensity training group. This prediction was tested with a linear mixed model, according to our statistical analysis plan; Test type: Superiority; p < .05, Mixed Models Analysis; Kenward-Roger adjustments for degrees of freedom; Slope = -0.02, 95% CI 2-sided [-.04 to .01] — Parameter is the interaction term for the interaction of group, learning rate, and session

2. Secondary Outcome: Change in Hippocampal-cortical Functional Connectivity
Description: The change in strength of the correlation between the spontaneous functional magnetic resonance imaging (fMRI) signal in the hippocampus and cortical regions in a hippocampal-cortical memory system.
Time Frame: Baseline, 30 minutes
Population: Before randomization in the parallel assignment intervention study, all participants completed an acute exercise manipulation that had a repeated measures, within-subject cross-over design for exposure to exercise intensity. Participants completed this acute exercise manipulation before randomization so participants are not yet in their chronic intervention arm. The N for each arm therefore corresponds to the n that was exposed to each of the acute exercise conditions.
Measure: Mean (Standard Error); unit: functional connectivity (correlation)
Groups:
- Moderate Intensity Aerobic Exercise; Light Intensity Aerobic Exercise: Acute manipulation
Arm/Group | Moderate Intensity Aerobic Exercise | Light Intensity Aerobic Exercise
Number analyzed (Participants) | 118 | 122
functional connectivity (correlation) | .001 (.005) | -.005 (.005)
Statistical Analysis 1: Comparison: Moderate Intensity Aerobic Exercise vs Light Intensity Aerobic Exercise; We tested the prediction that hippocampal-cortical functional connectivity would change more for the moderate-to-vigorous acute condition compared to the light intensity condition. This prediction was tested with a linear mixed model, according to our statistical analysis plan; Test type: Superiority; p < .05, Mixed Models Analysis; Kenward-Roger adjustments for degrees of freedom; Mean Difference (Final Values) = .01, 95% CI 2-sided [-.01 to .02] — Parameter is the interaction term for the interaction of exercise condition (intensity) and session

3. Secondary Outcome: Change in Hippocampal-cortical Functional Connectivity
Description: as for outcome 2
Time Frame: Baseline, 24-weeks
Measure: Mean (Standard Deviation); unit: functional connectivity (correlation)
Arm/Group | Cardiorespiratory Fitness Training | Functional Fitness Training
Number analyzed (Participants) | 50 | 48
functional connectivity (correlation) | -.007 (.07) | -.005 (.06)
Statistical Analysis 1: Comparison: Cardiorespiratory Fitness Training vs Functional Fitness Training; We tested the prediction that functional connectivity strength would increase more so for the moderate-to-vigorous training group compared to the light intensity training group. This prediction was tested with a linear mixed model, according to our statistical analysis plan; Test type: Superiority; p < .05, Mixed Models Analysis; Kenward-Roger adjustments for degrees of freedom; Mean Difference (Net) = 0, 95% CI 2-sided [-.03 to .02]; Parameter is the interaction term for the interaction of group and session

4. Secondary Outcome: Change in Cardiorespiratory Fitness
Description: Cardiorespiratory fitness will be measured during a maximal exercise test. Oxygen uptake (VO2) will be measured from expired air samples taken at 30 second intervals until a peak VO2, the highest VO2, is attained at the point of test termination due to symptom limitation and/or volitional exhaustion. Change in maximal VO2 is reported for descriptive results.
Time Frame: Baseline, 24-weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Cardiorespiratory Fitness Training | Functional Fitness Training
Number analyzed (Participants) | 48 | 44
ml/kg/min | 2.33 (2.26) | .53 (2.40)
Statistical Analysis 1: Comparison: Cardiorespiratory Fitness Training vs Functional Fitness Training; We tested the prediction that cardiorespiratory fitness would increase more so for the moderate-to-vigorous training group compared to the light intensity training group. This prediction was tested with a linear mixed model, as reported in our protocol paper; Test type: Superiority; p < .05, Mixed Models Analysis; Residualized change model, as reported in our protocol paper; Mean Difference (Final Values) = 1.42, 95% CI 2-sided [.27 to 2.59]

ADVERSE EVENTS:
Time Frame: The duration of enrollment for all participant, which includes from the time they signed informed consent until completion of their last post-intervention assessment. Typically this was 8 months.
Groups:
- Moderate Intensity Aerobic Exercise: Crossover condition of Moderate Intensity Aerobic Exercise preceding Light Intensity Aerobic Exercise for acute exercise manipulation
- Light Intensity Aerobic Exercise: Crossover condition of Light Intensity Aerobic Exercise preceding Moderate Intensity Aerobic Exercise for acute exercise manipulation
Arm/Group | Moderate Intensity Aerobic Exercise | Light Intensity Aerobic Exercise | Cardiorespiratory Fitness Training | Functional Fitness Training
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/122 | 0/60 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/122 | 0/60 | 0/56
Other Adverse Events (participants affected / at risk) | 0/119 | 0/122 | 22/60 | 8/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Intensity Aerobic Exercise (N=119) | Light Intensity Aerobic Exercise (N=122) | Cardiorespiratory Fitness Training (N=60) | Functional Fitness Training (N=56)
Pain (knee, joint, hip) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 16 (16) | 5 (5)
Heart abnormality at peak at fitness test (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Incidental finding in MRI (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Positive for COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT03114150/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2023-12-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT03114150/SAP_002.pdf